CLINICAL TRIAL: NCT00192231
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Investigate Immune Responses Elicited by a Liquid Formulation of Influenza Virus Vaccine, Trivalent Types A & B, Live Cold Adapted (CAIV-T) in Healthy Adults Aged 18 and Older
Brief Title: Trial to Investigate Immune Responses Elicited by a Liquid Formulation of Influenza Virus Vaccine,(CAIV-T)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D153 P510
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2006-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

INTERVENTIONS:
Biological: CAIV-T

SUMMARY:
The primary objective of this study was to perform a variety of immunological assays on blood, serum, nasal wash samples, and cells obtained from healthy adult subjects for the purpose of developing assays for application in the further investigation of immune responses generated by influenza virus vaccine, trivalent, types A and B, live, cold-adapted (liquid CAIV-T).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 59 years or > 60 years.
* Female subjects of childbearing potential who had a negative urine pregnancy test result prior to study vaccination. Females who were surgically sterilized or post-menopausal did not require pregnancy testing.
* Adults who were determined by medical history, physical examination and clinical judgment eligible for this study. Subjects with stable pre-existing disease, defined as disease not requiring change in therapy or hospitalization within 12 weeks before receipt of study vaccination, were eligible.
* Subjects who provided written informed consent after the nature of the study was explained.
* Subjects who were available for the duration of the study (from enrollment to study completion).
* Subjects who could be reached by study staff for the post-vaccination contact [via telephone, clinic or home visit].

Exclusion Criteria:

* Subjects who resided in a nursing home or long-term care facility or other institution receiving skilled or semi-skilled nursing care. An ambulatory subject who resided in a retirement home or village was eligible for participation.
* Subjects with evidence of dementia or other severe cognitive impairment based on Mini Mental State Examination (MMSE) score of 22 or greater. Note: Administration of MMSE was performed only if clinically indicated.

For all study subjects:

* Subjects who were perceived to be unavailable or difficult to contact for evaluation of study visits during the study period.
* Subjects with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids; or cytotoxic agents.
* Subjects who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study.
* Subjects who resided in the same household as an immunosuppressed or immunocompromised individual.
* Subjects with a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccine or placebo.
* Subjects who were administered any live virus vaccine within one month prior to enrollment.
* Subjects for whom there was intent to administer any other investigational vaccine or agent from one month prior to enrollment through the conclusion of the study.
* Subjects who received a dose of influenza treatment (commercial or investigational) one month prior to enrollment. Prophylactic use of influenza antivirals was not permitted.
* Subjects who received any influenza vaccine in the six months prior to enrollment, or nonstudy influenza vaccine since enrollment.
* Subjects with any medical conditions that in the opinion of the investigator might interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2001-04; Study Completion 2001-06

PRIMARY OUTCOMES:
The safety objective was to assess the safety and tolerability of CAIV-T vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (1):
- Austin & Repatriation Medical Centre, Heidelburg, Victoria, Australia